CLINICAL TRIAL: NCT06684847
Title: A Phase 3 Randomized, Double-Blinded, Placebo-Controlled Multicenter Trial With Open-Label Extension to Evaluate the Efficacy, Safety, and Tolerability of Efgartigimod PH20 Subcutaneous Administered by Prefilled Syringe in Adult Patients With Primary Sjögren's Disease
Brief Title: A Study of the Efficacy and Safety of Efgartigimod in Patients With Primary Sjögren's Syndrome
Acronym: Unity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2306; 2024-516609-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Primary Sjogrens Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blinded treatment period: Efgartigimod PH20 SC (Experimental): Participants receiving efgartigimod PH20 SC during the double-blinded treatment period
  Interventions: Biological: Efgartigimod PH20 SC
- Double-blinded treatment period: Placebo PH20 SC (Placebo Comparator): Participants receiving placebo PH20 SC during the double-blinded treatment period
  Interventions: Other: Placebo PH20 SC
- Open-label treatment period (Experimental): Participants receiving efgartigimod PH20 SC during the open-label treatment period
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — subcutaneous efgartigimod PH20 SC given by prefilled syringe
  Arms: Double-blinded treatment period: Efgartigimod PH20 SC; Open-label treatment period
Other: Placebo PH20 SC — subcutaneous placebo PH20 SC given by prefilled syringe
  Arms: Double-blinded treatment period: Placebo PH20 SC

SUMMARY:
The main purpose of the proposed study is to evaluate the efficacy of efgartigimod PH20 SC in patients with moderate-to-severe Primary Sjögren's Disease (pSjD). The study consists of a double-blinded placebo-controlled treatment period and an open-label treatment period. The maximum study duration for participants in both study parts is approximately 105 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies when signing the ICF.
* Meets the following criteria at screening: fulfilled ACR/EULAR classification criteria 2016 PSjD criteria before screening; clinESSDAI ≥ 6 at screening; Anti-Ro/SS-A positive at central laboratory; Unstimulated residual salivary flow (≥ 0.01 mL/min)

Exclusion Criteria:

* Secondary (also referred to as associated) Sjögren's disease, defined as overlap with another autoimmune rheumatic or systemic inflammatory condition (eg, rheumatoid arthritis, systemic lupus erythematosus, scleroderma, or idiopathic inflammatory myopathy
* Active fibromyalgia which is not adequately controlled in the judgment of the investigator, or participant is receiving fibromyalgia treatment that has not been stable treatment for at least 12 weeks before screening.
* Any severe systemic pSjD manifestation that is not adequately controlled at screening or baseline that may put the participant at undue risk based on the investigator's opinion.
* Use of cyclophosphamide ≤ 24 weeks prior to screening
* Anti-CD20 or anti-CD19 antibody received < 6 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in clinESSDAI score at week 48 | Up to 48 weeks
  The ESSDAI was designed to measure systemic disease activity in patients with PSjD and consists of 12 domains. The score varies between 0 (no disease activity) and 123 (max disease activity). The clinESSDAI includes all ESSDAI domains except the biological domain.

SECONDARY OUTCOMES:
Change from baseline in ESSDAI score at week 48 | Up to 48 weeks
  The ESSDAI was designed to measure systemic disease activity in patients with PSjD and consists of 12 domains. The score varies between 0 (no disease activity) and 123 (max disease activity).
Proportion of participants with low disease activity (clinESSDAI < 5) at week 48 | Up to 48 weeks
  The ESSDAI was designed to measure systemic disease activity in patients with PSjD and consists of 12 domains. The score varies between 0 (no disease activity) and 123 (max disease activity). The clinESSDAI includes all ESSDAI domains except the biological domain.
Proportion of responders on STAR (defined as ≥ 5 points) at week 48 | Up to 48 weeks
  Sjögren's Tool for Assessing Response ( STAR) has been developed as a composite score to assess the efficacy of treatments for PSjD in 5 domains. Patients are classified as STAR responders when they reach ≥ 5 of 9 points.
Change from baseline in DiSSA joint pain item at week 48 | Up to 48 weeks
  Diary of Sjögren's Symptoms Assessment (DiSSA) is a patient-reported symptom severity diary that includes 6 PSjD symptoms. Each symptom is rated from 0 (no symptoms) to 10 (worst).
Change from baseline in DiSSA total score at week 48 | Up to 48 weeks
  Diary of Sjögren's Symptoms Assessment (DiSSA) is a patient-reported symptom severity diary that includes 6 PSjD symptoms. Each symptom is rated from 0 (no symptoms) to 10 (worst).
Change from baseline in DiSSA sicca domain at week 48 | Up to 48 weeks
  Diary of Sjögren's Symptoms Assessment (DiSSA) is a patient-reported symptom severity diary that includes 6 PSjD symptoms. Each symptom is rated from 0 (no symptoms) to 10 (worst).
Proportion of participants with MCII (minimal clinically important improvement) in ESSDAI (defined as improvement of ≥ 3 points) at week 48 | Up to 48 weeks
  The ESSDAI was designed to measure systemic disease activity in patients with PSjD and consists of 12 domains. The score varies between 0 (no disease activity) and 123 (max disease activity).
Change from baseline in clinESSDAI score at week 24 | Up to 24 weeks
  The ESSDAI was designed to measure systemic disease activity in patients with PSjD and consists of 12 domains. The score varies between 0 (no disease activity) and 123 (max disease activity). The clinESSDAI includes all ESSDAI domains except the biological domain.

CONTACTS AND LOCATIONS:
Locations (276):
- United States (32):
  - One of a Kind Clinical Research Center LLC, Scottsdale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Tucson, Arizona
  - Providence Medical Foundation, Fullerton, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Life Clinical Trials, Margate, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - St. Luke's Clinic - Rheumatology, Boise, Idaho
  - Chicago Clinical Research Institute, Chicago, Illinois
  - Great Lakes Clinical Trials, LLC Ravenswood dba Flourish Research, Chicago, Illinois
  - Greater Chicago Specialty Physicians LLC, Orland Park, Illinois
  - Arizona Arthritis & Rheumatology Research, PLLC, Willowbrook, Illinois
  - Accurate Clinical Research Inc., Lake Charles, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Samaritan Health Services, Corvallis, Oregon
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Allen Arthritis, Allen, Texas
  - Accurate Clinical Management, Baytown, Texas
  - Novel Research LLC, Bellaire, Texas
  - Precision Comprehensive Clinical Research Solution, Colleyville, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Arizona Arthritis & Rheumatology Research, PLLC, Fort Worth, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - North Houston Arthritis Center, Houston, Texas
  - Arizona Arthritis & Rheumatology Research, PLLC, Irving, Texas
  - R and H Clinical Research, Katy, Texas
  - Simcare Medical Research LLC, Sugar Land, Texas
  - Velocity Clinical Research Waco, Waco, Texas
- Argentina (13):
  - Centro Medico Arsema, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Centro de Investigaciones San Miguel, San Miguel, Buenos Aires
  - Sanatorio Parque S.A., Rosario, Santa Fe Province
  - Instituto CAICI, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - STAT Research S.A., Buenos Aires
  - Centro Medico Barrio Parque, Buenos Aires
  - Consultorios Reumatologicos Pampa, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - APRILLUS Asistencia e Investigacion, Buenos Aires
- Australia (4):
  - Westmead Hospital, Sydney, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch
- Rheuma-Zentrum Wien Oberlaa, Vienna, Austria
- Belgium (5):
  - Erasme Hospital, Brussels
  - University Hospital Antwerp, Edegem
  - ReumaClinic, Genk
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Bulgaria (4):
  - MC Artmed OOD, Plovdiv
  - UMHAT "Pulmed" OOD, Plovdiv
  - MHAT Dr Ivan Seliminski AD, Sliven
  - DCC "Alexandrovska" EOOD, Sofia
- Canada (2):
  - Applied Medical Informatics Research Inc., Montreal, Quebec
  - G.R.M.O Groupe De Recherche En Maladie Osseuses Inc, Québec
- Chile (6):
  - CTR Estudios, Santiago
  - Enroll Spa, Santiago
  - BioMedica Research Group, Santiago
  - Centro de Estudios Reumatologicos, Santiago
  - Centro Medico Prosalud, Santiago
  - Clinical Research Chile SpA., Valdivia
- China (35):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi Zhuang
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Jining No.1 People's Hospital, Jining, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Linfen Central Hospital, Linfen, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Kunming Medical College Affiliated First Hospital, Kunming, Yun'Nan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
- Colombia (12):
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Barranquilla
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Clinica de la Costa S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - BlueCare S.A.S, Bogotá
  - Sociedad de Cirugia de Bogota Hospital de San Jose, Bogotá
  - Servimed S.A.S., Bucaramanga
  - IPS Centro Medico Julian Coronel S.A., Cali
  - Preventive Care Ltda, Chía
  - Hospital Pablo Tobon Uribe, Medellín
  - Servicios De Salud IPS Suramericana S A S IPS Sura Industriales Medellin, Medellín
  - Healthy Medical Center, Zipaquirá
- Estonia (3):
  - OÜ Innomedica, Tallinn
  - Center for Clinical and Basic Research, Tallinn
  - Meditrials, Tartu
- France (4):
  - Hôpital Saint Joseph, Marseille, Bouches-du-Rhône
  - CHR Orléans, Orléans, Loiret
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Georgia (7):
  - The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Geo Hospitals LLC, Tbilisi
  - VIAN, Tbilisi
  - MediClub Georgia LLC, Tbilisi
  - Clinic on Mtskheta Street, Tbilisi
  - First Medical Center, Tbilisi
  - Innova LLC, Tbilisi
- Germany (4):
  - Universitaetsklinikum, Tübingen, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen, Munich, Bavaria
  - HRF II - Hamburger Rheuma Forschungszentrum II, Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Greece (5):
  - Euroclinic of Athens, Athens
  - NNA Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - University General Hospital Attikon, Chaïdári
  - General Hospital Papageorgiou, Thessaloniki
- Hungary (5):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Bekes Varmegyei Kozponti Korhaz, Gyula
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Vita Verum Medical, Székesfehérvár
- Ireland (2):
  - Clinical Research Ctr, Dublin
  - Respiratory Depart Research, Dublin
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - The Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (3):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Stabilimento Ospedaliero Santa Chiara, Pisa
  - Università Campus Bio-Medico di Roma - UOC Reumatologia, Roma
- Japan (20):
  - JCHO Chukyo Hospital, Nagoya, Aichi-ken
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiya-shi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Sasebo Chuo Hospital, Sasebo-shi, Nagasaki
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Shimane University Hospital, Izumo-shi, Shimane
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - St. Luke's International Hospital, Chūōku, Tokyo-To
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - NHO Tokyo Medical Center, Meguro-ku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
- Jordan (6):
  - The Specialty Hospital Advanced Clinical Center, Amman
  - Jordan University Hospital, Amman
  - Abdali Hospital, Amman
  - Istiklal Hospital, Amman
  - Pharmaceutical research center at Jordan University of Science and Technology, Irbid
  - Irbid Specialty Hospital, Irbid
- Lebanon (4):
  - Saint George Hospital University Medical Center, Beirut
  - American University of Beirut, Beirut
  - Hotel Dieu de France Hospital, Beirut
  - Ain Wazein Medical Village, El Shouf
- Lithuania (3):
  - Siauliai Republican Hospital, Šiauliai
  - Inlita, JSC, Center of Santaros Clinical Trials, Vilnius
  - Vilnius University Hospital, Vilnius
- Mexico (13):
  - CIMAB SA de CV, Torreón, Coahuila
  - CIMOVA (Consultorio anexo), León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Panamerican Clinical Research Mexico S.A. de C.V. Guadalajara, Guadalajara, Jalisco
  - Centro de investigacion medica y reumatologia, Guadalajara, Jalisco
  - Consultorio Privado Dr. Miguel Cortes Hernandez, Cuernavaca, Morelos
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa SC, Culiacán, Sinaloa
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Medical Care & Research SA de CV, Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, Sociedad Civil, Chihuahua City
  - Centro de Investigacion y Atencion Integral Durango S.C., Durango
  - Clinstile, S.A. de C.V., Mexico City
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Philippines (4):
  - Ospital Ng Makati, City of Taguig
  - Manila Doctors Hospital, Manila
  - The Medical City, Ortigas
  - St. Luke's Medical Center, Quezon City
- Poland (32):
  - Nova Reuma, Bialystok
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Centrum Medyczne Intercor Sp. z o.o, Bydgoszcz
  - Centrum Medyczne K2J2, Częstochowa
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Ambulatorium Sp z o o, Elblag
  - FutureMeds Gdynia, Gdynia
  - MCBK Iwona Czajkowska Anna Podrażka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Centrum Medyczne Pratia Katowice, Katowice
  - Malopolskie Badania Kliniczne, Krakow
  - FutureMeds Krakow, Krakow
  - SOMED CR, Lodz
  - FutureMeds, Lodz
  - Clinical Trials Umed Sp.z o.o, Lodz
  - ETG Lublin, Lublin
  - Reumed Spolka z o.o., Lublin
  - Provita Profamilia, Piotrkow Trybunalski
  - Pratia Poznan, Poznan
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan
  - Clinical Research Center Spółka z, Poznan
  - ETG Siedlce, Siedlce
  - MICS Centrum Medyczne Warszawa, Warsaw
  - ETG JustMed, Warsaw
  - PRATIA S.A. MTZ Clinical Research Powered by Pratia, Warsaw
  - Izabela Inglot Szczebiot, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - FutureMeds, Warsaw
  - REUMA CENTRUM Specjalistyczna Praktyka Lekarska, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - FutureMeds, Wroclaw
  - ETG Zamosc, Zamość
- Portugal (3):
  - Unidade Local de Saude de Coimbra, Coimbra
  - Hospital CUF Descobertas, Lisbon
  - Hospital Conde de Bertiandos - Ponte de Lima (Unidade Local do Alto Minho, EPE), Ponte de Lima
- Romania (3):
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - S.C Delta Health Care S.R.L, Bucharest
  - SC Aqua Med Consulting SRL, Constanța
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Special Hospital for Rheumatic Diseases, Novi Sad
- Slovakia (5):
  - Artromac, Košice
  - MEDMAN s.r.o., Martin
  - MEDMAN, Martin
  - Narodny ustav reumatickych chorob, Piešťany
  - ALBAMED, Zvolen
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Soonchunhyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (11):
  - Hospital Universitario de Badajoz, Badajoz, Badajoz
  - Sanitas ES Sanitas Hospital CIMA, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron - VHIR, Barcelona, Barcelona
  - Clinica GAIAS Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid, Spain
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Studieenheten, Stockholm, Sweden
- Tunisia (4):
  - Hopital Habib Thameur, Montfleury
  - EPS Hopital Mohamed Taher Maamouri, Nabeul
  - Hedi Chaker Hospital, Sfax
  - Hospital Farhat Hached, Sousse
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- United Kingdom (3):
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Hallamshire Hospital, Sheffield, West Midlands
  - Cannock Chase Hospital, Cannock

IPD SHARING:
Plan to Share IPD: No